CLINICAL TRIAL: NCT01140347
Title: A Multicenter, Randomized, Double-Blind, Phase 3 Study of Ramucirumab (IMC-1121B) Drug Product and Best Supportive Care (BSC) Versus Placebo and BSC as Second-Line Treatment in Patients With Hepatocellular Carcinoma Following First-Line Therapy With Sorafenib (REACH)
Brief Title: A Study of Ramucirumab (IMC-1121B) Drug Product (DP) and Best Supportive Care (BSC) Versus Placebo and BSC as 2nd-Line Treatment in Participants With Hepatocellular Carcinoma After 1st-Line Therapy With Sorafenib
Acronym: REACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13895; CP12-0919 (Other: ImClone Systems); I4T-IE-JVBF (Other: Eli Lilly and Company); 2010-019318-26 (EudraCT Number)
Record Dates: First submitted 2010-06-02; First posted 2010-06-09 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma (HCC); recombinant human immunoglobulin G; subclass 1 (IgG1) monoclonal antibody (MAb); Hepatocellular Carcinoma (HCC) following First-Line Therapy With Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramucirumab DP and BSC (Experimental)
  Interventions: Biological: Ramucirumab DP (IMC-1121B); Other: BSC
- Placebo and BSC (Placebo Comparator)
  Interventions: Biological: Placebo; Other: BSC

INTERVENTIONS:
Biological: Placebo — 8 mg/kg IV every 2 weeks
  Arms: Placebo and BSC
Biological: Ramucirumab DP (IMC-1121B) — 8 milligrams/kilogram (mg/kg) intravenous (IV) every 2 weeks
  Other Names: IMC-1121B; LY3009806
  Arms: Ramucirumab DP and BSC
Other: BSC — Palliative and supportive care for disease-related symptoms and toxicity associated with treatment as deemed medically necessary and appropriate in the opinion of the investigator.

SUMMARY:
This is a Phase 3 multicenter, randomized study evaluating the safety and efficacy of ramucirumab DP plus BSC as a double-blind, placebo-controlled (placebo plus BSC) comparison.

Approximately 544 participants, at least 18 years of age, with Child-Pugh score < 7 and diagnosed with hepatocellular carcinoma will be randomized. Participants must have received sorafenib as first-line systemic treatment for hepatocellular carcinoma (HCC), and must have discontinued sorafenib prior to entering the study.

Hypothesis: This sample size will allow differentiation of the expected increase in median overall survival (OS), from 8 months in the placebo arm to 10.67 months in the ramucirumab arm.

Upon registration and completion of screening procedures, eligible participants with HCC who have disease progression during or following first-line therapy with sorafenib, or were intolerant to this agent, will be randomized to receive either ramucirumab DP or placebo.

The treatment regimen will be continued until radiographic or symptomatic progression, the development of unacceptable toxicity, noncompliance or withdrawal of consent by the participant, or investigator decision.

ELIGIBILITY:
Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Child-Pugh score of <7 (Child-Pugh Class A only)
* Barcelona Clinic Liver Cancer (BCLC) Stage C or BCLC stage B not amenable to locoregional therapy or refractory to locoregional therapy
* Diagnosis of HCC (excluding fibrolamellar carcinoma) in the absence of histologic or cytologic confirmation
* There are either clinical, laboratory, or radiographic findings consistent with a diagnosis of liver cirrhosis
* Has a liver mass measuring at least 2 centimeters (cm) with characteristic vascularization seen on either triphasic computed tomography (CT) scan or magnetic resonance imaging (MRI) with gadolinium
* At least 1 measurable or evaluable lesion that is viable [that is (i.e.), is vascularized], and has not been previously treated with locoregional therapy. A lesion that has been previously treated will qualify as a measurable or evaluable lesion if there was demonstrable progression following locoregional therapy
* Previously treated with sorafenib and has discontinued sorafenib treatment at least 14 days prior to randomization. Participants may have experienced:

  * Radiographically documented disease progression during sorafenib therapy or after discontinuation of sorafenib therapy, or
  * Discontinuation of sorafenib due to an adverse drug reaction, despite dose reduction by 1 level and BSC
* The participant has received sorafenib as the only systemic therapeutic intervention. Any hepatic locoregional therapy that has been administered prior to sorafenib is allowed, but not following sorafenib. Radiation to metastatic sites [for example (e.g.), bone] following sorafenib therapy is permitted.
* Resolution of clinically significant toxicity of any anti-cancer therapy to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events volume 4.0 (NCI-CTCAE v. 4.0).

Adequate Organ Function defined as:

* Total bilirubin <3.0 milligrams/deciliter (mg/dL) [51.3 micromole/liter (µmol/L)], aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × upper limit of normal (ULN)
* Serum creatinine ≤1.2 × ULN or calculated creatinine clearance >50 milliliters/minute (mL/min)
* Absolute neutrophil count (ANC) ≥1.0 × 10^3/microliter (μL) (1.0 × 10^9/liter (L)]), hemoglobin ≥9 grams/deciliter (g/dL) [5.58 millimoles/liter (mmol/L)], and platelets ≥75 × 10^3/µL (75 × 10^9/L)
* International Normalized Ratio (INR) ≤1.5 and partial thromboplastin time (PTT) ≤5 seconds above ULN. Participants receiving prophylactic low-dose anticoagulant therapy are eligible provided that INR ≤1.5 and PTT ≤5 seconds above the ULN
* The participant's urinary protein is ≤1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates ≥2+ proteinuria, then a 24-hour urine must be collected and must demonstrate <1000 milligrams (mg) of protein in 24 hours to allow participation in the study

Exclusion criteria:

* Major surgery within 28 days prior to randomization, or central venous access device placement within 7 days prior to randomization
* Hepatic locoregional therapy within 28 days prior to randomization
* Radiation to any nonhepatic (e.g., bone) site within 14 days prior to randomization
* Sorafenib within 14 days prior to randomization
* Received any investigational therapy or non-approved drug within 28 days prior to randomization
* Received any previous systemic therapy with vascular endothelial growth factor (VEGF) inhibitors or vascular endothelial growth factor receptor (VEGFR) inhibitors (including investigational agents) other than sorafenib for treatment of HCC
* Fibrolamellar carcinoma
* Received any transfusion, blood component preparation, erythropoietin, albumin preparation, or granulocyte colony-stimulating factors (G-CSF) within 14 days prior to randomization
* Therapeutic anticoagulation with warfarin, low-molecular-weight heparin, or similar agents. Participants receiving prophylactic, low-dose anticoagulation therapy are eligible provided that the coagulation parameters defined in the inclusion criteria (INR ≤1.5 and PTT ≤5 seconds above the ULN) are met
* Receiving ongoing therapy with nonsteroidal anti-inflammatory agents (NSAIDs, e.g., indomethacin, ibuprofen, naproxen, nimesulide, celecoxib, etoricoxib, or similar agents) or other antiplatelet agents (e.g., clopidogrel, ticlopidine, prasugrel, dipyridamole, picotamide, indobufen, anagrelide, triflusal). Aspirin (ASA) at doses up to 100 milligrams/day (mg/day) is permitted
* Symptomatic congestive heart failure, unstable angina pectoris, or symptomatic or poorly controlled cardiac arrhythmia
* Any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization
* Uncontrolled arterial hypertension systolic ≥150 / diastolic ≥90 millimeters of mercury (mm Hg) despite standard medical management
* Grade 3-4 gastrointestinal bleeding or any variceal bleeding episode in the 3 months prior to randomization requiring transfusion, endoscopic or operative intervention (participants with any bleeding episode considered life-threatening during the 3 months prior to randomization are excluded, regardless of transfusion or intervention status)
* Esophageal or gastric varices that require immediate intervention (e.g., banding, sclerotherapy) or represent a high bleeding risk. Participants with evidence of portal hypertension (including splenomegaly) or any prior history of variceal bleeding must have had endoscopic evaluation within the 3 months immediately prior to randomization. Participants with evidence of portal hypertension are eligible for study participation if endoscopic evaluation does not indicate esophageal or gastric varices that require immediate intervention or represent a high bleeding risk; however, these eligible participants must receive supportive therapy (e.g., beta blocker therapy) according to institutional standards and clinical guidelines during study participation
* Central nervous system (CNS) metastases or carcinomatous meningitis
* History of or current hepatic encephalopathy or current clinically meaningful ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (146):
- United States (18):
  - ImClone Investigational Site, Orange, California
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, New Haven, Connecticut
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, New Orleans, Louisiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Worcester, Massachusetts
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Newark, New Jersey
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Winston-Salem, North Carolina
  - ImClone Investigational Site, Dayton, Ohio
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Lubbock, Texas
  - ImClone Investigational Site, Seattle, Washington
  - ImClone Investigational Site, Milwaukee, Wisconsin
- Australia (5):
  - ImClone Investigational Site, Bankstown, New South Wales
  - ImClone Investigational Site, Kogarah, New South Wales
  - ImClone Investigational Site, Liverpool Bc, New South Wales
  - ImClone Investigational Site, Kurralta Park, South Australia
  - ImClone Investigational Site, Prahran, Victoria
- Austria (4):
  - ImClone Investigational Site, Linz
  - ImClone Investigational Site, Salzburg
  - ImClone Investigational Site, Steyr
  - ImClone Investigational Site, Vienna
- Belgium (7):
  - ImClone Investigational Site, Bonheiden
  - ImClone Investigational Site, Brussels
  - ImClone Investigational Site, Charleroi
  - ImClone Investigational Site, Edegem
  - ImClone Investigational Site, Leuven
  - ImClone Investigational Site, Liège
  - ImClone Investigational Site, Ottignies
- Brazil (10):
  - ImClone Investigational Site, Belo Horizonte
  - ImClone Investigational Site, Botucatu
  - ImClone Investigational Site, Brasília
  - ImClone Investigational Site, Campinas
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Ribeirão Preto
  - ImClone Investigational Site, Rio de Janeiro
  - ImClone Investigational Site, Salvador
  - ImClone Investigational Site, Sao Jose Rio Preto
  - ImClone Investigational Site, São Paulo
- Bulgaria (3):
  - ImClone Investigational Site, Plovdiv
  - ImClone Investigational Site, Sofia
  - ImClone Investigational Site, Varna
- ImClone Investigational Site, Ottawa, Ontario, Canada
- Czechia (4):
  - ImClone Investigational Site, Brib
  - ImClone Investigational Site, Hradec Králové
  - ImClone Investigational Site, Olomouc
  - ImClone Investigational Site, Prague
- ImClone Investigational Site, Helsinki, Finland
- France (14):
  - ImClone Investigational Site, Amiens
  - ImClone Investigational Site, Angers
  - ImClone Investigational Site, Avignon
  - ImClone Investigational Site, Besançon
  - ImClone Investigational Site, Bordeaux
  - ImClone Investigational Site, Clermont-Ferrand
  - ImClone Investigational Site, La Roche-sur-Yon
  - ImClone Investigational Site, Limoges
  - ImClone Investigational Site, Marseille
  - ImClone Investigational Site, Nice
  - ImClone Investigational Site, Paris
  - ImClone Investigational Site, Poitiers
  - ImClone Investigational Site, Reims
  - ImClone Investigational Site, Saint-Etienne
- Germany (17):
  - ImClone Investigational Site, Berlin
  - ImClone Investigational Site, Bielefeld
  - ImClone Investigational Site, Bonn
  - ImClone Investigational Site, Düsseldorf
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Frankfurt
  - ImClone Investigational Site, Freiburg im Breisgau
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Hanover
  - ImClone Investigational Site, Homburg
  - ImClone Investigational Site, Leipzig
  - ImClone Investigational Site, Magdeburg
  - ImClone Investigational Site, Munich
  - ImClone Investigational Site, Münster
  - ImClone Investigational Site, Tübingen
  - ImClone Investigational Site, Ulm
  - ImClone Investigational Site, Weiden
- Hong Kong (3):
  - ImClone Investigational Site, Kowloon
  - ImClone Investigational Site, Pokfulam
  - ImClone Investigational Site, Shatin
- ImClone Investigational Site, Budapest, Hungary
- Israel (3):
  - ImClone Investigational Site, Beersheba
  - ImClone Investigational Site, Petah Tikva
  - ImClone Investigational Site, Tel Aviv
- Italy (12):
  - ImClone Investigational Site, Bari
  - ImClone Investigational Site, Benevento
  - ImClone Investigational Site, Bologna
  - ImClone Investigational Site, Genova
  - ImClone Investigational Site, Lecce
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Modena
  - ImClone Investigational Site, Padua
  - ImClone Investigational Site, Palermo
  - ImClone Investigational Site, Pavia
  - ImClone Investigational Site, Rome
  - ImClone Investigational Site, Udine
- Japan (14):
  - ImClone Investigational Site, Chiba
  - ImClone Investigational Site, Fukuoka
  - ImClone Investigational Site, Hyōgo
  - ImClone Investigational Site, Ishikawa
  - ImClone Investigational Site, Kanagawa
  - ImClone Investigational Site, Kochi
  - ImClone Investigational Site, Kyoto
  - ImClone Investigational Site, Miyagi
  - ImClone Investigational Site, Osaka
  - ImClone Investigational Site, Osaka-Pref
  - ImClone Investigational Site, Saga
  - ImClone Investigational Site, Tochigi
  - ImClone Investigational Site, Tokushima
  - ImClone Investigational Site, Tokyo
- Netherlands (2):
  - ImClone Investigational Site, Amsterdam
  - ImClone Investigational Site, Rotterdam
- ImClone Investigational Site, Oslo, Norway
- ImClone Investigational Site, Quezon City, Philippines
- Portugal (2):
  - ImClone Investigational Site, Lisbon
  - ImClone Investigational Site, Santa Maria da Feira
- Romania (3):
  - ImClone Investigational Site, Bucharest
  - ImClone Investigational Site, Cluj-Napoca
  - ImClone Investigational Site, Craiova
- South Korea (4):
  - ImClone Investigational Site, Anyang
  - ImClone Investigational Site, Incheon
  - ImClone Investigational Site, Seodaemun-Gu
  - ImClone Investigational Site, Seoul
- Spain (5):
  - ImClone Investigational Site, Ávila
  - ImClone Investigational Site, Girona
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Ourense
  - ImClone Investigational Site, Valencia
- ImClone Investigational Site, Stockholm, Sweden
- ImClone Investigational Site, Bern, Switzerland
- Taiwan (7):
  - ImClone Investigational Site, Changhua
  - ImClone Investigational Site, Kuei Shan Hsiang
  - ImClone Investigational Site, Liouying/Tainan
  - ImClone Investigational Site, Niaosung
  - ImClone Investigational Site, Taichung
  - ImClone Investigational Site, Tainan
  - ImClone Investigational Site, Taipei
- Thailand (2):
  - ImClone Investigational Site, Bangkok
  - ImClone Investigational Site, Hat Yai

REFERENCES:
- [Derived] Llovet JM, Singal AG, Villanueva A, Finn RS, Kudo M, Galle PR, Ikeda M, Callies S, McGrath LM, Wang C, Abada P, Widau RC, Gonzalez-Gugel E, Zhu AX. Prognostic and Predictive Factors in Patients with Advanced HCC and Elevated Alpha-Fetoprotein Treated with Ramucirumab in Two Randomized Phase III Trials. Clin Cancer Res. 2022 Jun 1;28(11):2297-2305. doi: 10.1158/1078-0432.CCR-21-4000. PMID 35247922
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Zhu AX, Finn RS, Kang YK, Yen CJ, Galle PR, Llovet JM, Assenat E, Brandi G, Motomura K, Ohno I, Daniele B, Vogel A, Yamashita T, Hsu CH, Gerken G, Bilbruck J, Hsu Y, Liang K, Widau RC, Wang C, Abada P, Kudo M. Serum alpha-fetoprotein and clinical outcomes in patients with advanced hepatocellular carcinoma treated with ramucirumab. Br J Cancer. 2021 Apr;124(8):1388-1397. doi: 10.1038/s41416-021-01260-w. Epub 2021 Feb 3. PMID 33531690
- [Derived] Reig M, Galle PR, Kudo M, Finn R, Llovet JM, Metti AL, Schelman WR, Liang K, Wang C, Widau RC, Abada P, Zhu AX. Pattern of progression in advanced hepatocellular carcinoma treated with ramucirumab. Liver Int. 2021 Mar;41(3):598-607. doi: 10.1111/liv.14731. Epub 2020 Dec 5. PMID 33188713
- [Derived] Zhu AX, Nipp RD, Finn RS, Galle PR, Llovet JM, Blanc JF, Okusaka T, Chau I, Cella D, Girvan A, Gable J, Bowman L, Wang C, Hsu Y, Abada PB, Kudo M. Ramucirumab in the second-line for patients with hepatocellular carcinoma and elevated alpha-fetoprotein: patient-reported outcomes across two randomised clinical trials. ESMO Open. 2020 Aug;5(4):e000797. doi: 10.1136/esmoopen-2020-000797. PMID 32817068
- [Derived] Kudo M, Okusaka T, Motomura K, Ohno I, Morimoto M, Seo S, Wada Y, Sato S, Yamashita T, Furukawa M, Aramaki T, Nadano S, Ohkawa K, Fujii H, Kudo T, Furuse J, Takai H, Homma G, Yoshikawa R, Zhu AX. Ramucirumab after prior sorafenib in patients with advanced hepatocellular carcinoma and elevated alpha-fetoprotein: Japanese subgroup analysis of the REACH-2 trial. J Gastroenterol. 2020 Jun;55(6):627-639. doi: 10.1007/s00535-020-01668-w. Epub 2020 Feb 27. PMID 32107609
- [Derived] Arnold D, Fuchs CS, Tabernero J, Ohtsu A, Zhu AX, Garon EB, Mackey JR, Paz-Ares L, Baron AD, Okusaka T, Yoshino T, Yoon HH, Das M, Ferry D, Zhang Y, Lin Y, Binder P, Sashegyi A, Chau I. Meta-analysis of individual patient safety data from six randomized, placebo-controlled trials with the antiangiogenic VEGFR2-binding monoclonal antibody ramucirumab. Ann Oncol. 2017 Dec 1;28(12):2932-2942. doi: 10.1093/annonc/mdx514. PMID 28950290
- [Derived] Chau I, Peck-Radosavljevic M, Borg C, Malfertheiner P, Seitz JF, Park JO, Ryoo BY, Yen CJ, Kudo M, Poon R, Pastorelli D, Blanc JF, Chung HC, Baron AD, Okusaka T, Bowman L, Cui ZL, Girvan AC, Abada PB, Yang L, Zhu AX. Ramucirumab as second-line treatment in patients with advanced hepatocellular carcinoma following first-line therapy with sorafenib: Patient-focused outcome results from the randomised phase III REACH study. Eur J Cancer. 2017 Aug;81:17-25. doi: 10.1016/j.ejca.2017.05.001. Epub 2017 Jun 4. PMID 28591675
- [Derived] Zhu AX, Baron AD, Malfertheiner P, Kudo M, Kawazoe S, Pezet D, Weissinger F, Brandi G, Barone CA, Okusaka T, Wada Y, Park JO, Ryoo BY, Cho JY, Chung HC, Li CP, Yen CJ, Lee KD, Chang SC, Yang L, Abada PB, Chau I. Ramucirumab as Second-Line Treatment in Patients With Advanced Hepatocellular Carcinoma: Analysis of REACH Trial Results by Child-Pugh Score. JAMA Oncol. 2017 Feb 1;3(2):235-243. doi: 10.1001/jamaoncol.2016.4115. PMID 27657674
- [Derived] Kudo M, Hatano E, Ohkawa S, Fujii H, Masumoto A, Furuse J, Wada Y, Ishii H, Obi S, Kaneko S, Kawazoe S, Yokosuka O, Ikeda M, Ukai K, Morita S, Tsuji A, Kudo T, Shimada M, Osaki Y, Tateishi R, Sugiyama G, Abada PB, Yang L, Okusaka T, Zhu AX. Ramucirumab as second-line treatment in patients with advanced hepatocellular carcinoma: Japanese subgroup analysis of the REACH trial. J Gastroenterol. 2017 Apr;52(4):494-503. doi: 10.1007/s00535-016-1247-4. Epub 2016 Aug 22. PMID 27549242
- [Derived] Zhu AX, Park JO, Ryoo BY, Yen CJ, Poon R, Pastorelli D, Blanc JF, Chung HC, Baron AD, Pfiffer TE, Okusaka T, Kubackova K, Trojan J, Sastre J, Chau I, Chang SC, Abada PB, Yang L, Schwartz JD, Kudo M; REACH Trial Investigators. Ramucirumab versus placebo as second-line treatment in patients with advanced hepatocellular carcinoma following first-line therapy with sorafenib (REACH): a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2015 Jul;16(7):859-70. doi: 10.1016/S1470-2045(15)00050-9. Epub 2015 Jun 18. PMID 26095784

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died due to any cause or were alive and on study at conclusion but off treatment were considered to have completed the study.
Groups:
- Ramucirumab (IMC-1121B) + BSC: Ramucirumab (IMC-1121B): 8 milligrams/kilogram (mg/kg) intravenous (IV) infusion every 2 weeks.
  Best supportive care (BSC): Palliative and supportive care for disease-related symptoms and toxicity associated with treatment as deemed medically necessary and appropriate in the opinion of the investigator.
- Placebo + BSC: Placebo: 8 mg/kg IV infusion every 2 weeks. BSC: Palliative and supportive care for disease-related symptoms and toxicity associated with treatment as deemed medically necessary and appropriate in the opinion of the investigator.
Period: Overall Study
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Started | 283 | 282
Received at Least 1 Dose of Study Drug | 277 | 276
Completed | 265 | 268
Not Completed | 18 | 14
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 13 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab (IMC-1121B) + BSC: Ramucirumab 8 mg/kg IV infusion every 2 weeks. BSC: Palliative and supportive care for disease-related symptoms and toxicity associated with treatment as deemed medically necessary and appropriate in the opinion of the investigator.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC | Total
Number analyzed (Participants) | 283 | 282 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.56) | 62.5 (11.10) | 62.7 (11.33)
Age, Customized [Number; unit: participants]
  <65 years | 150 | 162 | 312
  ≥65 years | 133 | 120 | 253
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 87
  Male | 236 | 242 | 478
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 253 | 260 | 513
  Unknown or Not Reported | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 131 | 135 | 266
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 139 | 137 | 276
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 37
  Portugal | 0 | 2 | 2
  Philippines | 1 | 0 | 1
  Taiwan | 33 | 25 | 58
  Hong Kong | 14 | 10 | 24
  Spain | 9 | 12 | 21
  Thailand | 5 | 1 | 6
  Israel | 1 | 1 | 2
  Switzerland | 1 | 1 | 2
  Italy | 33 | 18 | 51
  France | 32 | 27 | 59
  Australia | 3 | 8 | 11
  Netherlands | 2 | 1 | 3
  Korea, Republic of | 28 | 42 | 70
  Finland | 0 | 3 | 3
  Austria | 4 | 4 | 8
  Czech Republic | 11 | 9 | 20
  Hungary | 1 | 0 | 1
  Canada | 0 | 1 | 1
  Belgium | 3 | 5 | 8
  Brazil | 15 | 12 | 27
  Romania | 3 | 4 | 7
  Bulgaria | 2 | 4 | 6
  Germany | 19 | 21 | 40
  Norway | 1 | 1 | 2
  Japan | 45 | 48 | 93
  Sweden | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. Participants who were alive at the end of the follow-up period or were lost to follow-up were censored on the last date the participant was known to be alive.
Time Frame: Randomization to death from any cause (up to 37 months)
Population: Intent-to-treat (ITT) Population: All randomized participants. Participants censored: Ramucirumab+BSC (Ram)=65, Placebo+BSC (Pl)=58.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 283 | 282
months | 9.17 [8.05 to 10.64] | 7.62 [6.01 to 9.33]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + BSC vs Placebo + BSC; Test type: Superiority or Other; p = 0.1391, Log Rank; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.717 to 1.046] — HR with 95% confidence interval (CI) was estimated using a stratified Cox proportional hazards regression model using the Interactive Web Response System (IWRS) stratification factors (geographical regions and etiology of liver disease)

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from date of randomization until date of objectively determined progressive disease (PD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 or death from any cause. PD was defined as ≥20% increase in sum of diameters (SOD) of target lesions, taking as reference smallest sum on study (including baseline sum if it was smallest). Sum must show a ≥5 millimeter (mm) increase. Appearance of ≥1 new lesions and unequivocal progression of existing non-target lesions were considered progression. In primary analysis, participants alive and without PD were censored at day of last adequate tumor assessment; progression or deaths without progression occurring immediately after ≥2 missed tumor assessments, were censored at day of the last adequate tumor assessment prior to missing assessments; participants who began new anticancer therapy were censored at day of the last adequate tumor assessment prior to start of new anticancer therapy.
Time Frame: Randomization to PD (up to 36 months)
Population: ITT Population: All randomized participants. Participants censored: Ram=43, Pl=19.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 283 | 282
months | 2.79 [2.69 to 3.94] | 2.10 [1.58 to 2.69]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + BSC vs Placebo + BSC; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.625, 95% CI 2-sided [0.522 to 0.750] — HR with 95% CI was estimated using a stratified Cox proportional hazards regression model using the IWRS stratification factors (geographical regions and etiology of liver disease)

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: ORR was defined, using RECIST v1.1 criteria, as the percentage of participants who achieved a best overall response of CR or PR. CR was defined as the disappearance of all lesions and any intratumor arterial enhancement in target lesions, the normalization of the tumor marker level and all lymph nodes short axis reduced to <10 mm. PR was defined as ≥30% decrease in the SOD of target lesions, including the short axes of any target lymph nodes, taking as reference the baseline SOD of target lesions, no new lesions and stable nontarget lesions. Percentage of participants was calculated as: (number of participants with CR or PR / number of participants randomized) * 100.
Time Frame: Baseline to the date of first evidence of confirmed CR or PR (up to 37 months)
Population: ITT Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 283 | 282
percentage of participants | 7.1 [4.6 to 10.7] | 0.7 [0.2 to 2.5]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + BSC vs Placebo + BSC; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) adjusted for geographic region and etiology liver disease

4. Secondary Outcome: Time to Radiographic Progression (TTP)
Description: TTP was defined as the time from randomization to the first radiographically documented PD. PD was defined, using RECIST v1.1 criteria, as ≥20% increase in SOD of target lesions, taking as reference smallest sum on study (including baseline sum if it was the smallest). Sum must show an absolute increase of ≥5 mm. Appearance of ≥1 new lesions and unequivocal progression of existing non-target lesions were considered progression. Participants without PD were censored at the day of the last adequate tumor assessment. Progression occurred immediately after ≥2 missed tumor assessments and were censored at the day of the last adequate tumor assessment prior to the missing assessments. Participants who began new anticancer therapy were censored at the day of their last adequate tumor assessment prior to start of new anticancer therapy.
Time Frame: Randomization to PD (up to 36 months)
Population: ITT Population: All randomized participants. Participants censored: Ram=86, Pl=52.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 283 | 282
months | 3.48 [2.76 to 4.47] | 2.63 [1.58 to 2.76]
Statistical Analysis 1: Comparison: Ramucirumab (IMC-1121B) + BSC vs Placebo + BSC; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.593, 95% CI 2-sided [0.487 to 0.722] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy (FACT) Hepatobiliary Symptom Index-8 (FHSI-8)
Description: The FHSI-8 is a self-administered 8-item questionnaire that measures a participant's symptoms in the domains of jaundice, stomach pain/discomfort weight loss, and fatigue. Participants rated each item on a 5-point scale from 0 (not at all) to 4 (very much). Item scores were calculated as outlined in the FACIT manual. FHSI-8 total score was the sum of each item's score with a total score ranging from 0 (highly symptomatic) to 32 (asymptomatic).
Time Frame: Baseline, Prior to infusion on Day 1 of Cycle 4, Cycle 10, and Cycle 16 (14-day cycles), and end of treatment (up to 34 months)
Population: Randomized participants who had FHSI-8 at baseline and the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 169 | 199
units on a scale
  Cycle 4 (n=166, 147) | -1.26 (3.164) | -0.81 (4.623)
  Cycle 10 (n=70, 45) | -1.28 (3.989) | -0.01 (4.378)
  Cycle 16 (n=47, 24) | -0.97 (4.095) | 0.75 (3.768)
  End of Treatment (n=169, 199) | -2.44 (5.561) | -2.86 (5.618)

6. Secondary Outcome: Change From Baseline in European Quality of Life Questionnaire-5 Dimensions (EQ-5D) Health State Score
Description: The EQ-5D is a self-reported, 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire related to the participant's current health state. Each question was scored using a 3 level scale (no problems, some problems, or extreme problems). EQ-5D health state was defined by combining responses from each of the 5 dimensions into a weighted health-state index score according to the United Kingdom (UK) population based algorithm where 0 = death and 1 = perfect health.
Time Frame: Baseline, Prior to infusion on Day 1 of Cycle 4, Cycle 10, and Cycle 16 (14-day cycles), end of treatment (up to 34 months)
Population: Randomized participants who had an EQ-5D score at baseline and the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 166 | 190
units on a scale
  Cycle 4 (n=166, 145) | -0.038 (0.189) | -0.046 (0.245)
  Cycle 10 (n=71, 45) | -0.054 (0.212) | 0.003 (0.148)
  Cycle 16 (n=47, 25) | -0.062 (0.214) | -0.012 (0.085)
  End of Treatment (n=166, 190) | -0.129 (0.290) | -0.144 (0.280)

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and the Number of Participants Who Died
Description: The number of participants with serious AEs (SAEs), other non-serious AEs and participants who died. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (up to 37 months)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 276
participants
  SAEs | 123 | 92
  Other Non-SAEs | 254 | 235
  Died | 215 | 220

8. Secondary Outcome: Maximum Concentration (Cmax) of Ramucirumab, Cycle 1
Time Frame: 1 hour following the completion of Cycle 1 (14-day cycle) infusion
Population: Participants who received Cycle 1 of Ram and had Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ramucirumab (IMC-1121B) + BSC
Number analyzed (Participants) | 247
micrograms/milliliter (µg/mL) | 149.6 (36.9)

9. Secondary Outcome: Cmax of Ramucirumab, Cycle 4
Time Frame: 1 hour following completion of Cycle 4 (14-day cycles) infusion
Population: Participants who received Cycle 4 of Ram and had Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1121B) + BSC
Number analyzed (Participants) | 140
µg/mL | 189.5 (39.1)

10. Secondary Outcome: Cmax of Ramucirumab, Cycle 7
Time Frame: 1 hour following completion of Cycle 7 (14-day cycles) infusion
Population: Participants who received Cycle 7 of Ram and had Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ramucirumab (IMC-1121B) + BSC
Number analyzed (Participants) | 81
µg/mL | 184.4 (56.3)

11. Secondary Outcome: Number of Participants With Treatment Emergent Positive Anti-Ramucirumab Response [Serum Anti-Ramucirumab Antibody Assessment (Immunogenicity)]
Description: Participants were considered positive for anti-ramucirumab antibodies [anti-drug antibodies (ADA)] if the post-treatment sample had an increase of at least 4-fold in titer from the pretreatment values. If the pretreatment value was not detected or was not present, a 1:20 post-treatment titer was required to indicate treatment emergence of ADA.
Time Frame: Prior to treatment and 1 hour post end of infusion for Cycles 1, 4 and 7 (14-day cycles)
Population: Participants who received at least 1 dose of study drug and had post-treatment ADA analysis.
Measure: Number; unit: participants
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Number analyzed (Participants) | 241 | 231
participants | 10 | 7

ADVERSE EVENTS:
Arm/Group | Ramucirumab (IMC-1121B) + BSC | Placebo + BSC
Serious Adverse Events (participants affected / at risk) | 124/277 | 92/276
Other Adverse Events (participants affected / at risk) | 254/277 | 235/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) + BSC (N=277) | Placebo + BSC (N=276)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 8 (8) | 3 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 (5) | 10 (12)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 4 (5) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 9 (9) | 3 (4)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 3 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (2) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 5 (8) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 6 (9) | 5 (9)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 4 (4) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 3 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (4)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (30) | 16 (22)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Coma hepatic (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 12 (16) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Tongue biting (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (4) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (4) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) + BSC (N=277) | Placebo + BSC (N=276)
Anaemia (Blood and lymphatic system disorders) | 29 (54) | 31 (44)
Leukopenia (Blood and lymphatic system disorders) | 14 (54) | 7 (19)
Neutropenia (Blood and lymphatic system disorders) | 16 (80) | 4 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 48 (189) | 12 (26)
Abdominal distension (Gastrointestinal disorders) | 19 (27) | 28 (31)
Abdominal pain (Gastrointestinal disorders) | 45 (63) | 58 (86)
Abdominal pain upper (Gastrointestinal disorders) | 26 (34) | 25 (32)
Ascites (Gastrointestinal disorders) | 72 (110) | 40 (47)
Constipation (Gastrointestinal disorders) | 36 (39) | 34 (39)
Diarrhoea (Gastrointestinal disorders) | 50 (74) | 38 (52)
Gingival bleeding (Gastrointestinal disorders) | 18 (22) | 4 (4)
Nausea (Gastrointestinal disorders) | 52 (71) | 52 (74)
Vomiting (Gastrointestinal disorders) | 30 (39) | 40 (47)
Asthenia (General disorders) | 50 (80) | 36 (63)
Fatigue (General disorders) | 66 (97) | 60 (99)
Oedema peripheral (General disorders) | 100 (151) | 50 (58)
Pyrexia (General disorders) | 42 (59) | 25 (32)
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 (16) | 15 (32)
Nasopharyngitis (Infections and infestations) | 15 (15) | 14 (16)
Alanine aminotransferase increased (Investigations) | 13 (34) | 21 (33)
Aspartate aminotransferase increased (Investigations) | 30 (59) | 39 (70)
Blood alkaline phosphatase increased (Investigations) | 18 (40) | 14 (25)
Blood bilirubin increased (Investigations) | 19 (39) | 24 (38)
Decreased appetite (Metabolism and nutrition disorders) | 59 (81) | 50 (62)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 (66) | 14 (27)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (21) | 15 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (26) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (27) | 23 (32)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 (26) | 12 (13)
Dizziness (Nervous system disorders) | 23 (25) | 16 (18)
Headache (Nervous system disorders) | 53 (69) | 15 (18)
Insomnia (Psychiatric disorders) | 19 (20) | 20 (20)
Proteinuria (Renal and urinary disorders) | 46 (117) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (54) | 25 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (33) | 26 (33)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (48) | 17 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (17) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (33) | 29 (41)
Rash (Skin and subcutaneous tissue disorders) | 23 (27) | 12 (16)
Hypertension (Vascular disorders) | 55 (104) | 20 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.